CLINICAL TRIAL: NCT00931320
Title: Investigation Into the RAtio of LDL-CHolestEroL to HDL-Cholesterol Improvement After Statin Treatment in Korean Patients
Acronym: RACHEL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Hyunah Caroline, Choi / CV TA Physician, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CKR-DUM-2009/3
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Dyslipidemias
Keywords: Ratio improvement; LDL-C; HDL-C; Ratio of Low Density Lipoprotein Cholesterol to High Density Lipoprotein Cholesterol Improvement; High Density Lipoprotein Cholesterol
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3000 patients: Who have at least made 1 visit to the outpatient clinic within previous 6 months .

SUMMARY:
An observational, non-interventional, multi-centre study to provide further information on the ratio of LDL-C to HDL-C improvement after statin treatment in Korean patients group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are taking lipid-lowering medication after diagnosed as dyslipidaemia
* Subjects who have at least made 1 visit to the outpatient clinic within previous 6 months
* Subjects who have records of both LDL-C and HDL-C before & after statin treatment (at least four weeks after statin taking)

Exclusion Criteria:

* Subjects who are unwilling or unable to provide their examination and lab result of medical chart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Who have at least made 1 visit to the outpatient clinic within previous 6 months .
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-07; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Evaluate current LDL/HDL ratio in Korean patients (between baseline & after treatment) | After Treatment : at least 4 weeks before statin taking /Baseline : no limitation.

SECONDARY OUTCOMES:
Evaluate difference of LDL/HDL ratio among different statins & dosages (between baseline & after treatment) | After Treatment : at least 4 weeks before statin taking / Baseline : no limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Hyunah Caroline Choi, Study Director — AstraZeneca Korea